CLINICAL TRIAL: NCT03723772
Title: A Trial Investigating the Pharmacokinetics and Pharmacodynamics of NNC0148-0287 C (Insulin 287) at Steady State Conditions in Subjects With Type 1 Diabetes
Brief Title: A Research Study of How Different Doses of a New Medicine NNC0148-0287 C (Insulin 287) Work on the Blood Sugar in People With Type 1 Diabetes When it is Taken Once a Week
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4225; U1111-1204-8909 (Other: World Health Organization (WHO)); 2017-004528-31 (EudraCT Number)
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin 287 followed by insulin glargine U100 (Experimental): Run-in period (2 days to 4 weeks): The basal insulin glargine dose for each subject will be established and optimised.
  After run-in, participants will receive insulin 287 once a week (OW) for 8 weeks and subsequent 4 weeks of terminal pharmacokinetic sampling where subjects are treated with once daily (OD) insulin glargine.
  After insulin 287 treatment, participants will receive insulin glargine U100 OD for 2 weeks.
  Interventions: Drug: Insulin icodec; Drug: IGlar U100
- Insulin glargine U100 followed by insulin 287 (Experimental): Run-in period (2 days to 4 weeks): The basal insulin glargine dose for each subject will be established and optimised.
  After run-in, participants will receive insulin glargine U100 OD for 2 weeks followed by 1-14 days (at least 1 day is mandatory) of continued insulin glargine treatment.
  After insulin glargine treatment, participants will receive insulin 287 once a week (OW) for 8 weeks and subsequent 4 weeks of terminal pharmacokinetic sampling.
  Interventions: Drug: Insulin icodec; Drug: IGlar U100

INTERVENTIONS:
Drug: Insulin icodec — Participants will receive subcutaneous injections of insulin 287 once weekly for 8 weeks
  Other Names: Insulin 287
Drug: IGlar U100 — Participants will receive subcutaneous injections of insulin glargine once weekly for 2 weeks.

SUMMARY:
This study compares the new long-acting insulin 287 with the marketed insulin glargine for use in type 1 diabetes. The study will test how insulin is taken up in your blood, how long it stays there and how the blood sugar is lowered. The participant will get both of the insulins in a random order. Insulin 287 is a new medicine while insulin glargine is already approved for the treatment of diabetes and can be prescribed by a doctor. The participant will get 8 weekly doses of insulin 287 and 14 daily doses of insulin glargine. There will also be a run-in period of 2 days to 4 weeks with daily doses of insulin glargine before you start the insulin 287 period. All doses will be injected under the skin. The study will last for about 16 to 24 weeks. The participant will have 27 visits with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-64 years (both inclusive) at the time of signing informed consent
* Diagnosed with type 1 diabetes mellitus greater than or equal to 1 year prior to the day of screening
* Current daily basal insulin treatment greater than or equal to 0.2 U/kg/day
* Body mass index between 18.5 and 29.0 kg/m^2 (both inclusive)
* HbA1c less than or equal to 9.0%

Exclusion Criteria:

* History or presence of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal or endocrinological conditions. Subjects with complications associated to diabetes can be included only if they are judged to be mild by the investigator. Subjects with other comorbidities (e.g. dyslipidaemia, hypertension and hypothyroidism) can be included if they have a stable treatment and are in adequate control according to the judgement of the investigator- Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice)
* Known or suspected hypersensitivity to trial products or related products

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
AUCI287,τ,SS - Area under the serum insulin 287 concentration-time curve during one dosing interval at steady state | From 0 to 168 hours after trial product administration (Day 50)
  Measured in pmol*h/L

SECONDARY OUTCOMES:
AUCGIR,16-52h,SS (for insulin 287) - Area under the glucose infusion rate-time curve at steady state | From 16 to 52 hours after trial product administration (Day 50)
  Measured in mg/kg
AUCGIR,138-168h,SS (for insulin 287) - Area under the glucose infusion rate-time curve at steady state | From 138 to 168 hours after trial product administration (Day 50)
  Measured in mg/kg
GIRmax,16-52h, SS (for insulin 287) - Maximum observed glucose infusion rate at steady state | From 16 to 52 hours after trial product administration (Day 50)
  Measured in mg/(kg*min)
GIRmax,138-168h, SS (for insulin 287) - Maximum observed glucose infusion rate at steady state | From 138 to 168 hours after trial product administration (Day 50)
  Measured in mg/(kg*min)
AUCGIR,0-24h,SS (for insulin glargine) - Area under the glucose infusion rate-time curve at steady state | From 0 to 24 hours after trial product administration (Day 14)
  Measured in mg/kg
GIRmax,0-24h, SS (for insulin glargine) - Maximum observed glucose infusion rate at steady state | From 0 to 24 hours after trial product administration (Day 14)
  Measured in mg/(kg*min)
AUCI287,0-168h,FD (from insulin 287) - Area under the serum insulin 287 concentration-time curve after the first dose | From 0 to 168 hours after trial product administration (Day 1)
  Measured in pmol*h/L
Cmax,I287,FD (for insulin 287) - Maximum observed serum insulin 287 concentration after the first dose | From 0 to 168 hours after trial product administration (Day 1)
  Measured in pmol/L
tmax,I287,FD (for insulin 287) - Time to maximum observed serum insulin 287 concentration after the first dose | From 0 to 168 hours after trial product administration (Day 1)
  Measured in hours
Cmax,I287,SS (for insulin 287) - Maximum observed serum insulin 287 concentration after the last dose | From 0 to 168 hours after trial product administration (Day 50)
  Measured in pmol/L
tmax,I287,SS (for insulin 287) - Time to maximum observed serum insulin 287 concentration after the last dose | From 0 to 168 hours after trial product administration (Day 50)
  Measured in hours
t½,I287,SS (for insulin 287) - Terminal half-life for insulin 287 at steady state | Terminal part of the serum insulin 287 concentration-time curve where the curve is well approximated by a straight line on logarithmic scale after last trial product administration (Day 50)
  Measured in hours
CI287,trough (for insulin 287) - Serum insulin 287 trough concentration | Measured at the end of each dosing interval 168 hours after trial product administration (Day 8, 15, 22, 29, 36, 43, 50 and 57)
  Measured in pmol/L
AUCIGlar,τ,SS (for insulin glargine) - Area under the serum insulin glargine concentration-time curve during one dosing interval at steady state | From 0 to 24 hours after trial product administration (Day 14)
  Measured in pmol*h/L
Cmax,IGlar,SS (for insulin glargine) - Maximum observed serum insulin glargine concentration at steady state | From 0 to 24 hours after trial product administration (Day 14)
  Measured in pmol/L
tmax,IGlar,SS (for insulin glargine) - Time to maximum observed serum insulin glargine concentration at steady state | From 0 to 24 hours after trial product administration (Day 14)
  Measured in hours
CIGlar,trough (for insulin glargine) - Serum insulin glargine trough concentration | Measured at the end of each dosing interval 24 hours after trial product administration (Day 4, 7, 14 and 15)
  Measured in pmol/L
Number of adverse events (AEs) | From first trial product administration (Day 1) to end of last dosing interval (Day 57 for insulin 287, day 15 for IGlar)
  Number of events
Number of hypoglycaemic episodes | From first trial product administration (Day 1) to end of last dosing interval (Day 57 for insulin 287, day 15 for IGlar)
  Number of episodes
Change in anti-insulin 287 antibody level | From first insulin 287 administration (Day 1) to Follow-up visit (visit 25, day 106)
  Measured in % B/T (percentage of bound tracer measured after precipitation to total tracer)
Change in anti-insulin 287 antibody titres | From first insulin 287 administration (Day 1) to Follow-up visit (visit 25, day 106)
  Number of dilutions
Positive cross-reactive anti-human insulin antibodies | At the follow-up visit (Visit 25, day 106)
  Number of patients with/without positive cross-reactive anti-human insulin antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Hovelmann U, Engberg S, Heise T, Kristensen NR, Norgreen L, Zijlstra E, Ribel-Madsen R. Pharmacokinetic and pharmacodynamic properties of once-weekly insulin icodec in individuals with type 1 diabetes. Diabetes Obes Metab. 2024 May;26(5):1941-1949. doi: 10.1111/dom.15510. Epub 2024 Feb 20. PMID 38379002